CLINICAL TRIAL: NCT07235072
Title: Comparative Analysis of Passive Fit and Time Efficiency in Allon-X Implants Protocols Using Photogrammetry, Splinted Scan Bodies, and Conventional Impression Technique
Brief Title: Passive Fit and Time Efficiency in All On-X Implants Protocols Using Photogrammetry, Splinted Scan Bodies, and Conventional Impression Technique
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Mohammed Fathy Abdelhamid, Master's Degree Candidate , Prosthodontics Department, October 6 University, October 6 University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: RECO6U/22-2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Passive Fit of Full-arch Implant Prostheses

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Photogrammetry-Based Full-Arch Impression (Experimental)
  Interventions: Device: Photogrammetry-Based Full-Arch Impression
- Digital Impression Using Splinted Scan Bodies (Experimental)
  Interventions: Device: Digital Impression Using Splinted Scan Bodies
- Conventional Open-Tray Implant Impression (Active Comparator)
  Interventions: Procedure: Conventional Open-Tray Implant Impression

INTERVENTIONS:
Device: Photogrammetry-Based Full-Arch Impression — Use of a photogrammetry system to capture the positions of All-on-X implants digitally without physical impression materials. The technique aims to achieve precise passive fit and reduce chairside working time. Measurements of passive fit discrepancy and total procedure time will be recorded
  Arms: Photogrammetry-Based Full-Arch Impression
Device: Digital Impression Using Splinted Scan Bodies — Digital full-arch impression using splinted scan bodies connected with resin to enhance stability. An intraoral scanner captures the splinted assembly for framework fabrication. Passive fit and working time will be evaluated
  Arms: Digital Impression Using Splinted Scan Bodies
Procedure: Conventional Open-Tray Implant Impression — Traditional full-arch open-tray impression using polyether or VPS material with splinted impression copings. This serves as the standard comparator for evaluating passive fit and procedure duration
  Arms: Conventional Open-Tray Implant Impression

SUMMARY:
compare the passive fit of three impression techniques: photogrammetry, intraoral digital scanning with splinted scan bodies, and the conventional open-tray impression technique, within the context of the All-on-X treatment concept. This comparison is expected to provide valuable clinical evidence to support clinicians in making informed decisions when considering the adoption of digital alternatives to conventional methods.

DETAILED DESCRIPTION:
For edentulous patients undergoing full-arch rehabilitation, the All-on-X treatment approach has proven to be a very successful option, providing enhanced function, aesthetics, and patient satisfaction. Achieving passive fit, which reduces mechanical stress on implants and prosthetic components and reduces the possibility of problems such screw loosening, fracture, or marginal bone loss, is crucial to the long-term effectiveness of implant-supported prostheses. Passive fit has traditionally been evaluated after prostheses are fabricated using traditional open-tray impression techniques, which are regarded as the gold standard because of their great precision and dependability. These approaches, however, are challenging, technique-specific, and susceptible to human mistake or material deformation. Other methods include digital intraoral scanning with splinted scan bodies and photogrammetry have become more appreciated due to the quick development of digital dentistry. Potential advantages of these digital workflows include quicker digital data transfer to the lab, less chairside time, and improved patient comfort. In the context of the All-on-X procedure, there is still no clinical data comparing the accuracy especially passive fit and time efficiency of these more recent methods with traditional impressions, despite these benefits. Thus, the purpose of this study is to compare the time efficiency and passive fit of three impression techniques: traditional open-tray impressions, digital intraoral scanning with splinted scan bodies, and photogrammetry. The findings will provide clinicians with evidence-based insights into whether digital alternatives can match or surpass traditional techniques in terms of accuracy and workflow efficiency, ultimately supporting the transition toward more modern, streamlined protocols in implant prosthodontics.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 45-65 years.

Fully edentulous or partially edentulous maxilla requiring full-arch rehabilitation.

Sufficient maxillary bone volume to support at least four implants according to the All-on-X protocol.

Systemically healthy patients with no contraindications to dental implant surgery (ASA I-II classification).

Demonstrated ability to maintain adequate oral hygiene.

Willingness to participate in the study and comply with follow-up visits and required maintenance protocols.

Patients seeking a fixed, implant-supported prosthesis for the maxilla due to missing teeth and inability to use removable prostheses effectively.

Acceptable radiographic findings with no signs of pathology, infection, or significant anatomical limitations.

Exclusion Criteria:

Uncontrolled systemic diseases (e.g., uncontrolled diabetes, osteoporosis, immunosuppressive disorders)

History of radiation therapy to the head and neck region

Active periodontal disease or untreated caries

Maxillary cysts, tumors, or pathologies

Poor oral hygiene or inability to maintain postoperative care

Insufficient bone volume for All-on-X without extensive grafting

Maxillary sinus pathology or oroantral fistula

Psychiatric illness or cognitive impairment affecting compliance

Bruxism or parafunctional habits

Pregnant or lactating women

History of implant failure or titanium allergy

Use of bisphosphonates or antiresorptive medications

Heavy smoking (>10 cigarettes/day)

Inability or unwillingness to attend follow-up visits

Diagnosed or symptomatic temporomandibular joint disorders (pain, clicking, locking, limited opening)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Passive fit measured using 3D inspection software (Geomagic Control X) | Immediately after framework verification

SECONDARY OUTCOMES:
Time efficiency, assessed using stop watch and measured by seconds. | During impression procedure

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Jasim AG, Abo Elezz MG, Altonbary GY, Elsyad MA. Accuracy of digital and conventional implant-level impression techniques for maxillary full-arch screw-retained prosthesis: A crossover randomized trial. Clin Implant Dent Relat Res. 2024 Aug;26(4):714-723. doi: 10.1111/cid.13336. Epub 2024 May 10. PMID 38727015
- [Result] Papaspyridakos P, De Souza A, Finkelman M, Sicilia E, Gotsis S, Chen YW, Vazouras K, Chochlidakis K. Digital vs Conventional Full-Arch Implant Impressions: A Retrospective Analysis of 36 Edentulous Jaws. J Prosthodont. 2023 Apr;32(4):325-330. doi: 10.1111/jopr.13536. Epub 2022 May 31. PMID 35524647
- [Result] Drancourt N, Auduc C, Mouget A, Mouminoux J, Auroy P, Veyrune JL, El Osta N, Nicolas E. Accuracy of Conventional and Digital Impressions for Full-Arch Implant-Supported Prostheses: An In Vitro Study. J Pers Med. 2023 May 15;13(5):832. doi: 10.3390/jpm13050832. PMID 37241002

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT07235072/Prot_SAP_000.pdf